CLINICAL TRIAL: NCT02289573
Title: Effects of NAVA and PSV to AECOPD Patients' Air Distribution and Dead Space
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Southeast University, China (Other)
Responsible Party: Principal Investigator, Jianfeng Xie, MD, Southeast University, China
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2014ZDSYLL086.0
Record Dates: First submitted 2014-10-16; First posted 2014-11-13 (Estimated); Last update posted 2014-11-13 (Estimated); Status verified 2014-10

CONDITIONS: Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- neurally adjusted ventilatory assist (Experimental)
  Interventions: Device: NAVA and PSV
- pressure support ventilation (Sham Comparator)
  Interventions: Device: NAVA and PSV

INTERVENTIONS:
Device: NAVA and PSV — change ventilation modes(NAVA and PSV) with different support levels

SUMMARY:
Chronic obstructive pulmonary disease(COPD) is a common disease among people. Acute exacerbation of chronic obstructive pulmonary disease(AECOPD) is the acute and aggravating phase of COPD which may lead to respiratory failure. Mechanical ventilation is a very important therapy for those patients,but traditional ventilation modes have some defects, so investigators need to find new modes to solve these problems. In this study, the investigators compare neurally adjusted ventilatory assist (NAVA) and PSV to observe the effects on AECOPD patients' air distribution and dead space to determine if NAVA is a more appropriate ventilation mode for AECOPD patients.

ELIGIBILITY:
Inclusion Criteria:

* AECOPD patients who need invasive mechanical ventilation
* Patients who can tolerate assist mechanical ventilation
* Patients who have signed ICF

Exclusion Criteria:

* Patients who are younger than 18 years old or older than 75 years old
* Patients whose respiratory center is severely inhibited
* Patients who can not stand NAVA gastric tube
* Patients who have coagulation disorders
* Patients whose vital signs are unstable
* Patients who are in other clinical trails

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2014-11; Primary Completion 2015-06 (Estimated); Study Completion 2015-06 (Estimated)

PRIMARY OUTCOMES:
the ratio of physiologic dead space over tidal volume (VD/VT) | 1 year

REFERENCES:
- [Derived] Sun Q, Liu L, Pan C, Zhao Z, Xu J, Liu A, Qiu H. Effects of neurally adjusted ventilatory assist on air distribution and dead space in patients with acute exacerbation of chronic obstructive pulmonary disease. Crit Care. 2017 Jun 2;21(1):126. doi: 10.1186/s13054-017-1714-1. PMID 28578708